CLINICAL TRIAL: NCT01581060
Title: A Phase I/II, Open-label, Dose-escalation Study to Investigate the Safety, Pharmacokinetics, Pharmacodynamics and Clinical Activity of the MEK Inhibitor WX-554 in Patients With Solid Tumours
Brief Title: Phase I/II Dose-escalation Study to Investigate Safety and Pharmacokinetics/ Pharmacodynamics of WX-554 in Patients With Solid Tumours
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study terminated for business reasons
Sponsor: Heidelberg Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WX/80-003; 2011-003408-19 (EudraCT Number)
Record Dates: First submitted 2012-03-28; First posted 2012-04-19 (Estimated); Last update posted 2014-05-16 (Estimated); Status verified 2014-05

CONDITIONS: Advanced Solid Tumours

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- WX-554 (Experimental)
  Interventions: Drug: WX-554

INTERVENTIONS:
Drug: WX-554 — Capsules of WX-554

SUMMARY:
The aim of part 1 of this study is to determine the optimal biological dose (OBD) and maximum tolerated dose (MTD) for WX-554 and the recommended dose/dose schedules for the chronic treatment in part 2. The aim of part 2 is to further determine the safety and tolerability of chronic treatment with WX-554.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with advanced, metastatic and/or progressive solid tumours for whom there is no effective standard therapy available.
2. Evaluable or measurable disease
3. Has normal organ functions; is no greater than 2 on the ECOG Performance Scale
4. life expectancy of >3 months
5. negative hCG test in women of childbearing potential

Exclusion Criteria:

1. Patients who received an investigational anti-cancer drug within 4 weeks of starting the study
2. Patients who received major surgery, radiotherapy, or immunotherapy within 4 weeks of starting the study
3. Clinically significant, unresolved toxicity from previous anti-cancer therapy Patients
4. Patients who previously received a MEK inhibitor
5. Presence of active gastrointestinal disease or other condition that will interfere significantly with the absorption, distribution, metabolism, or excretion of drugs.
6. Known medical history of retinal vein occlusion, intraocular pressure greater than 21 mm Hg or patient considered at risk of retinal vein thrombosis.
7. Known HIV positivity or active hepatitis B or C infection.
8. History of clinically significant cardiac condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2012-03; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Part 1: Determination of the Optimal Biological Dose (OBD) by the assessment of ERK phosphorylation (pERK) in peripheral blood mononuclear cells (PBMC) and assessment of TNF-alpha in plasma. | Cycle 1 (21 days)
Part 1: Determination of the Maximum Tolerated Dose (MTD) for WX-554 by the evaluation of DLTs in 3-6 patients at the end of 1 treatment cycle | Cycle 1 (21 days)
Part 2: To further determine the safety and tolerability by evaluating the incidence and severity of adverse events and serious adverse events (as per CTCAE grading), changes in hematology and chemistry values, vital signs, ECGs. | expected average of 3-6 months

SECONDARY OUTCOMES:
Assessment of PK variables maximum observed concentration (Cmax), minimum observed concentration (Cmin), time at which Cmax was present (tmax), Area Under Curve (AUC) | PK profile on day 1 and day 8
Assessment of ERK phosphorylation (pERK) in PBMC and tissue, assessment of TNF-alpha in plasma after oral intake of the OBD/MTD. | expected average of 3-6 months
Tumour response evaluation using RECIST 1.1 | expected average of 3-6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Plummer, MD, Principal Investigator — Sir Bobby Robson Cancer Trials Research Centre
Locations (5):
- United Kingdom (5):
  - Queen's University Belfast Cancer Centre, Belfast
  - Beatson West of Scotland Cancer Centre, Glasgow
  - St James' Institute of Oncology, Leeds
  - Christie NHS Foundation Trust, Oak Road Treatment Centre, Manchester
  - Sir Bobby Robson Cancer Trials Research Centre, Newcastle upon Tyne